CLINICAL TRIAL: NCT05390554
Title: Effect of Buteyko Breathing Technique on Asthma Severity Control Among School-Age Children
Brief Title: Using Buteyko Breathing Technique to Control Asthma in School-Age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pediatric Asthma
Record Dates: First submitted 2022-03-21; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-04

CONDITIONS: Childhood Asthma
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Buteyko Breathing Technique (Experimental): single group pre-post test
  Interventions: Behavioral: Buteyko Breathing Technique

INTERVENTIONS:
Behavioral: Buteyko Breathing Technique — * The child was instructed to sit and take a relaxed posture in a vertical chair, relax his shoulders and lean his lower back against the back of the chair.
  * Until conducting CP, the child was told to avoid alternate breathing, the child was asked to take a small breath in (two seconds), a small breath out (three seconds) and clutch the nose with empty lungs but not too clear on the 'out-breath. To prevent air from escaping through the airways, clutching the nose is necessary.
  * The researcher estimates how many seconds the child can continue safely before the need to breathe in again,
  * The child was told to hold their breath until the first need to breathe in was felt. Release the nose then and naturally breathe through it smoothly.
  * The first intake of breath after the CP should be no higher than the breath before taking the measurement; the child should not hold the breath for too long as this could lead the child to take a major breath after measuring the CP.
  Other Names: Breathing Exercises

SUMMARY:
Asthma is a complex condition that can impair not only the child's physical growth but also his optimal functional capacity and performance. Buteyko Breathing Technique (BBT) is an exercise designed to regulate the breathing process. The Buteyko technique also proposes lifestyle changes beyond breathing, including diet, allergy avoidance, and stress control. This study aims to evaluate the effect of the Buteyko breathing technique on asthma severity control among school-age children. In Egypt, this technique was applied through five studies, four among adult patients and only one among children. At Mansoura University, only one study was conducted among adult patients, and no studies were conducted among children. To fulfill this knowledge gap, it is necessary to study the effect of this technique on asthma severity control among school-age children. This study will use the Childhood Asthma Control, Peak Expiratory Flow Rate, and Control Pause tests to evaluate the children's asthma severity control.

DETAILED DESCRIPTION:
Methods

Research design:

A quasi-experimental design, one group pre and post-test will be used to conduct this study.

Study setting:

The study will be conducted at the out-patient clinics of Mansoura University Children Hospital (MUCH), which provides health services to children cases from the Dakhlia governorate and Delta region as asthmatic children routinely come to follow up on their condition with their parents.

Subjects:

The sample size cannot be calculated as there is no specific annual statistical report about the admitted asthma condition to the sensitivity clinic, so a convenient sample of asthmatic school-age children who fulfills the following criteria through the data collection period (3 month) will be recruited.

Ethical considerations:

* Ethical approval will be obtained from the Research Ethics Committee. Then official permission will be obtained from the hospital administrative authority to collect data and conduct the study.
* Participants and their parents will be informed that participation in this study is voluntary, and they have the right to accept or refuse participation in the study. Written informed consent will be obtained from the children and their parents, who will accept to participate in the study after providing them with a complete and detailed description of the study including the purpose and benefits. Participants will be informed that their personal data will be kept confidential. All information taken from participants will be protected.

Data collection tools: Data will be collected using the following three tools.

I. Tool one; Structured interview sheet for children and their mothers.

It consisted of two parts as follow:

* Part one; school age child's Biodemographic and clinical data This part was developed by the researcher after reviewing relevant literatures (Chen, et al, 2016; Kuti, & Omole, 2017), and modifications of study supervisors.
* Part two; Childhood Asthma Control Test(C-ACT)

II. Tool two; Peak Expiratory Flow Rate (PEFR) test

Steps of PEFR assessment:

- Determining the percentage of PEFR, which equals: [PEFR% = (measured PEFR \ Predicted PEFR) ×100].

- The predicted PEFR will be calculated using the child's height by the following formula: [Predicted average PEF [L/min] = (Body height [cm] x 5.3) - 433] (Kopač, 2017).

* The actual PEFR will be estimated by:

  1. Each child will be studied in the direct sitting posture.
  2. The disposable mouthpiece will be calibrated to the peak flow meter mouthpiece.
  3. The pointer will be shifted to zero.
  4. The child will be told to maintain (horizontally) the level of the peak flow meter and to keep his fingers away from the pointer.
  5. The child will be asked to take a deep breath and tightly close his lips around the plastic disposable mouthpiece.
  6. The child will be ordered to puff as much as possible.
  7. The child will be told to note that it is determined by the velocity of his puff.
  8. The readings will be taken.
  9. The pointer will be shifted to zero again.
  10. This will be replicated three times by each child, and the highest reading will be recorded. ( American Lung Association 2019).

      III. Tool three; Control Pause Test (CP) adopted from Buteyko Clinic International (2014).
* Evaluating the Control Pause Breathing test using the following steps:

  1. The child will be instructed to sit and take a relaxed posture in a vertical chair, relax his shoulders and lean his lower back against the back of the chair.
  2. Until conducting CP, the child will be told to avoid alternate breathing; the child will be asked to take a small breath in (two seconds), a small breath out (three seconds), and clutch the nose with empty lungs but not too clear on the 'out-breath. To prevent air from escaping through the airways, clutching the nose is necessary.
  3. The researcher will estimate how many seconds the child can continue safely before breathing in again,
  4. The child will be told to hold their breath until the first need to breathe in is felt.
  5. The first intake of breath after the CP should be no higher than the breath before taking the measurement; the child should not hold the breath for too long as this could lead the child to take a major breath after measuring the CP.

Study intervention:

A. The preparatory phase:

* A learning booklet and a story will be prepared by the researcher in a simple Arabic language to meet the mother's needs and motivate the children after reviewing the articles and literature. The data collection instrument (children's peak flow meter with the number of disposable plastic mouthpieces, measuring tape, weight scale, stopwatch, disinfectant alcohol, and pen) will be prepared by the researcher.
* The content validity of the study tools will be assessed and revised by a jury that involved a panel of five experts in the Faculty of Nursing at Mansoura University. The tool will be revised for clarity, relevancy, applicability, comprehensiveness, understanding, and easiness for implementation, and modifications will be made according to their opinions. The content reliability of the study tools will be tested by using Cronbach's alpha test.

B. Exploratory phase:

1. Pilot study A pilot study will be carried out on four cases to evaluate the clarity, feasibility, and applicability of the study tools, educational booklet, and story. In addition, identifying the possible obstacles that might hinder data collection and overcoming it. These subjects won't be included in the study sample.
2. Fieldwork

   * Data collection will be extended over three months; the researcher will attend two days per week in the allergy outpatient clinic from 9.00 am to 2.00 pm, and each child will take the Buteyko educational program over four weeks, one session each week.
   * Before the intervention: at the first-week session (1-W):

     1- An individualized interview with the children and the caregiver will be conducted at the beginning of the first-week session, where the parent will sign the informed consent. Then All the study tools (C-ACT, PEFR, and CPT) will be assessed before the intervention to determine the baseline data.
   * During the intervention: at first, second, third, and fourth-week sessions (1-W, 2-W, 3-W, 4-W):

     1. Demonstrating Buteyko Breathing Technique (BBT) until the child adequately understands its steps. Starting with the steps of the first-week session then, adding the newly learned steps of each following week accordingly (1-W, 1+2-W, 1+2+3-W, 1+2+3+4-W) as follows:

        Week one exercise:
        * Starting with nose breathing
        * Relaxed breathing technique
        * The control pause technique
        * Advising of an hour of taping
        * Daily nose-breathing walk technique
        * Managing medication instruction
        * Buteyko education about how to stop cough

        Week two exercise
        * Extended pause technique
        * How to avoid colds and flu
        * Reduced breathing technique
        * Night-time nose breathing instruction

        Week three and four
        * Very reduced breathing technique
        * Lifestyle, diet, and sleep modification
     2. Evaluating the BBTpractice of the children and their parents. The child will be asked to redemonstrate the Buteyko steps until he has well-practiced them. They will be instructed to practice this technique at home regularly. Parents will also be instructed to help their children to practice twelve repetitions of the Buteyko steps per day: four repetitions in the morning, four repetitions in the afternoon, and four repetitions in the evening, and to record the number of steps done by their children in their Buteyko Steps Diary. Finally, they will be instructed to follow the modified lifestyle.
     3. Following each weekly BBT- educational session, each child will be Evaluated for PEFR and CPT to follow up on the child's prognosis (2-W, 3-W).
   * After the intervention: at the fourth-week session (4-W):

     1. At the end of the final session, the child will be evaluated for C-ACT, PEFR, and CPT to evaluate the post-test.

ELIGIBILITY:
Inclusion Criteria:

* The school age child of both sex whose age range from 6: 12 years to insure the ability of the child to perform Buteyko exercise.
* The child whose condition is mild to moderate as confirmed by the medical practitioner.
* The child treated from asthma only by medications and no other alternative treatment as revealed by their primary caregiver.
* The child and their parents not take any previous instruction about Buteyko method.
* The child and their parents were accepting participation for four weeks during the study.

Exclusion Criteria:

* The child who not have the inclusion criteria.
* The child with severe asthma, cardiac disease, mental retardation, pneumonia, infectious disease, lung disease, physical disabilities and psychiatric disorders as confirmed by the medical practitioner.
* The child who receive any other alternative therapy. The sample size was limited because the starting of the COVID 19 pandemic which affect the children attendance to the clinic and refusal from mothers to continue in the study program.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Childhood Asthma Control Test(C-ACT) | 4 weeks
  The tool is a valid test established by GlaxoSmithKline that involves seven questions to evaluate asthma control and the effects of asthma on diurnal activities among school age children. It has seven questions; the first four are answered by the children and the last three by their parents. Each question had four answer options for children, and six answer options for parents. This part completed at the first and final sessions as a pre and posttest.
  Its scores were categorized as the following:
  * 20:27 good asthma control
  * 10:19 moderate asthma control
  * Less than 10 poorly asthma control

SECONDARY OUTCOMES:
Peak Expiratory Flow Rate (PEFR) | 4 weeks
  The Peak Expiratory Flow Rate (PEFR) is person's maximum speed of expiration. It is measured with a mini wright peak flow meter device to display person's capability to expire out air through the bronchi. Therefore, it gives an understanding of the extent of obstruction in the airway. The predicted PEFR was calculated and compared with the actual value to determine the level of airway obstruction. Its interpretations are often categorized into three zones of depth; green, yellow, and red
  * Green zone: The peak flow result is between 80-100% of the child's predicted value. This is the clear zone.
  * Yellow zone: Peak flow result is between 50-79% of the child's predicted value. This is the caution zone.
  * Red zone: Peak flow result is less than 50% of the child's predicted value. This is an asthma crisis.
Control Pause Test (CP) | 4 weeks
  It was established by Dr. Buteyko to assess the depth of breathing and consequent retention of carbon dioxide, resultant oxygenation and health by using special breathing holding manner. This acts as a natural peak flow meter and it was used as diagnostic and therapeutic technique as it one of the major techniques of BBT.
  The scoring was categorized as follow:
  * Less than 10: health is severely affected.
  * 10 to less than 20: patient probably suffering from a chronic illness, along with symptoms, such as blocked nose, snoring, insomnia, coughing, short breath, asthma.
  * 20 to less than 40: most symptoms are not there, but may occur following a triggering event.
  * 40 and more: good health.

CONTACTS AND LOCATIONS:
Overall Officials: Fawzia E Abusaad, Professsor, Study Chair — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Background] Chen E, Shalowitz MU, Story RE, Ehrlich KB, Levine CS, Hayen R, Leigh AK, Miller GE. Dimensions of Socioeconomic Status and Childhood Asthma Outcomes: Evidence for Distinct Behavioral and Biological Associations. Psychosom Med. 2016 Nov-Dec;78(9):1043-1052. doi: 10.1097/PSY.0000000000000392. PMID 27749682
- [Background] Kuti BP, Omole KO. Epidemiology, triggers, and severity of childhood asthma in Ilesa, Nigeria: Implications for management and control. Niger Med J. 2017 Jan-Feb;58(1):13-20. doi: 10.4103/0300-1652.218412. PMID 29238123
- [Background] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Background] American Academy of Allergy Asthma and Immunology (AAAAI) (2019). New study sheds light on the challenges and barriers of severe asthma management available at: https://www.aaaai.org/About/News/News/asthma.
- [Background] Buteyko Clinic International (2014). Breathing Exercise 1: The Control Pause (Part I). Available at https://buteykoclinic.com/breathing-exercise-1-the-control-pause-part-i/
- [Background] Kopač, M. (2017). Calculation of Predicted Peak Expiratory Flow in Children with a Formula. Open J Asthma, 1(1), 007-008. Available at https://www.peertechz.com/articles/OJA-1-102.php